CLINICAL TRIAL: NCT04965779
Title: The Effect of Abdominal Binder Use on Postpartum Pain, Bleeding, and Breastfeeding Success in Women Who Undergo Cesarean Delivery
Brief Title: The Effect of Abdominal Binder Use on Postpartum Pain, Bleeding, and Breastfeeding Success in Cesarean Delivery Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Kara Pınar, Research Asisstant, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CukurovaUniversity_PK_01
Record Dates: First submitted 2021-06-18; First posted 2021-07-16 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Cesarean Section
Keywords: Cesarean Section; Pain; Bleeding; Breast Feeding; Abdominal binder; Nursing postpartum care
MeSH Terms: conditions — Pain; Hemorrhage; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Abdominal binder) (Experimental): The abdominal binder is applied after the women come to the clinic (postpartum 1st hour) following cesarean delivery and removed after the postpartum 48th hour. Postpartum nursing care in line with a follow-up protocol that was created based on the Republic of Turkey Ministry of Health's Postpartum Care Management Guide (2018) is provided together with the application of the abdominal binder.
  Interventions: Device: Abdominal Binder; Other: Postpartum nursing care
- Control group (No abdominal binder) (Active Comparator): Only postpartum nursing care in line with a follow-up protocol that was created based on the Republic of Turkey Ministry of Health's Postpartum Care Management Guide (2018) is provided with no abdominal binder or similar application.
  Interventions: Other: Postpartum nursing care

INTERVENTIONS:
Device: Abdominal Binder — Women in the intervention group use an abdominal binder from postpartum hour 1 to 48, and will be checked every 6 hours. The abdominal circumference of the women is measured at the anterior superior iliac spine and umbilicus level with a tape measure before the application, and the binder size is adjusted to be 5% smaller (approximately 0.5-1 cm) than the measurement obtained.
  Arms: Intervention group (Abdominal binder)
Other: Postpartum nursing care — Postpartum nursing care the follow-up protocol includes the evaluation and record between postpartum 1. and 48. hours of pain level, analgesic administration, follow-up of the puerperal bleeding, and uterine tone, measure of hemodynamic parameters measuring, hemoglobin level and hematocrit ratio, and assessment breastfeeding.

SUMMARY:
The aim of this randomized controlled interventional study is to identify the effect of the use of an abdominal binder on postpartum pain, bleeding, and breastfeeding success in primiparous women who have undergone planned cesarean delivery with spinal anesthesia.

DETAILED DESCRIPTION:
A 2015 report by the World Health Organization (WHO) has emphasized that cesarean section can be effective in preventing maternal and perinatal mortality and morbidity when there is a life-threatening danger to the mother and/or fetus, but provides no benefit to the woman or the baby otherwise. It also states that the ideal cesarean section rate 10% to 15%, and a rate above 10% at the population level is ineffective in decreasing maternal and infant mortality. However, current cesarean rates are much higher than recommended, especially in developed western countries, and rates ranging from 14.8% (Israel) to 54.8% (Turkey) have been reported as of 2018. Turkey, with a rate of 54.8%, has the highest cesarean section rate among the reported data.

Cesarean delivery is common worldwide and presents many maternal and neonatal risks. While bleeding is the most serious of these risks, the women also experience severe pain and face problems with breastfeeding. The risk of a postpartum bleeding complication is reported to be 2.5 times higher in women who have undergone a planned cesarean section. The rate of experiencing any pain after a cesarean section has been reported as 77% to 92.7% while the incidence of moderate/severe pain is 15.2% to 52.2%. In addition, the probability of experiencing breastfeeding problems in the post-cesarean period is reported to be approximately 7 times higher.

The need for optimum care in the postpartum period in order to protect the health of both the mother and the newborn, and also to prevent the health problems that may develop in the short and long term has been emphasized. Appropriate interventions of the nurses who are in close contact with the women, the newborns, and the families during the postpartum period affect the quality of care significantly. Based on this information, the various effects of the post-cesarean use of an abdominal binder, which is a noninvasive nursing intervention, has been evaluated in the literature and shown to have various benefits in the management of postpartum complications and problems after cesarean section in women with various characteristics. A limited number of studies have reported that the use of an abdominal binder decreases pain but inconsistent effect on postpartum bleeding. However, there is no study evaluating the effect of abdominal binder use on breastfeeding success.

The study was planned as a randomized controlled interventional study with the women randomly divided into intervention (abdominal binder) and control groups. A preliminary application was used to determine the sample size of the study. Based on the power analysis performed with the data obtained, a total of 128 women were included in the study with 64 women in each group, at a confidence interval of 95%, power of 90%, and α level of 0.05.

Block random sampling method was adopted to recruit participants. In order to randomly assign the participants to the groups, a list of 1:1 random numbers was created with the software Research Randomizer (https://www.randomizer.org/) on the computer. Participants were assigned to groups by 8-block randomization method. Randomization was done by an expert statistical consultant who was not responsible for conducting the study. The determined randomization number of list was printed out separately and sealed in each envelope. The random number was hidden in sealed envelopes until participants approved to participate in the study. Writing the random numbers on the papers, placing them in the envelopes and opening the paper in the sealed envelopes were done by an independent volunteer who was not responsible for the conduct of the study. Those who meet the inclusion and exclusion criteria and approve to participate in the study was allocated to intervention (abdominal binder) group or control group according to the result of randomization. In order to prevent bias each participant in the groups was followed in different rooms from the other participants in the group to which they were assigned.

SPSS software (IBM Corp., Armonk, NY, v. 24.0) will be used to evaluate the data. Descriptive analysis will be calculated using mean and standard deviation, median and interquartile range for continuous variables, and percentage and frequency for categorical variables. Independent sample t-tests, Mann-Whitney U test, chi-square test or Fisher's exact test will be used to compare any differences in socio-demographic data or outcome variables between groups. To determine the differences or changes between study group and control group (between group effects), within group effects (time), and the interaction effects (group x time), repeated measures analysis of variances (RM-ANOVA) and to compare the variables with two repeated measurements paired sample t-test will be applied when assumptions for parametric test are fulfilled. When the data cannot fulfill the assumptions of parametric test, Mann-Whitney U test will be applied to compare the differences between groups at each time interval while Friedman test will be used to determine the time effects within each group. Significant results are indicated if p-value of all statistical analysis is less than 0.05 for two-tailed test.

Tools for measuring the outcome variables in this study have been demonstrated validity and reliability (Breastfeeding Assesment Scale [LATCH]) and selectivity (Visual Analog Scale [VAS]) in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Can read and write in Turkish,
* Conscious and cooperating,
* Aged ≥19 to <35 years,
* At the ≥38th gestational week,
* Primiparous,
* With a healthy, singleton pregnancy and fetus,
* Scheduled to undergo cesarean delivery under spinal anesthesia and then undergoes the procedure,
* A minimum blood hemoglobin level of ≥11 g/dl and minimum hematocrit ratio of ≥36% at the time of cesarean delivery,
* Has the infant with her from cesarean delivery until discharge

Exclusion Criteria:

* A maternal systemic disease,
* A chronic pain problem or regular use of pain medications,
* A psychiatric disease,
* Scheduled to undergo or has undergone any intervention or drug administration in the pre-/intra-/post-operative period,
* Development of any complication in the pre-/intra-/post-operative period,
* Drain placement in the postpartum period

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — At the ≥38th gestational week
Enrollment: 128 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Postpartum pain evaluation for cesarean section incision | Since postpartum arrival to the clinic (postpartum hour 1) up to 48 hours
  Postpartum pain level evaluation for cesarean section incision in this study is determined using Visual Analog Scale [VAS]. VAS is a self-report tool used in the subjective assessment of pain. It is in the form of a 10 cm (100 mm) ruler with no pain at one end (minimum pain score=0) and the most severe pain at the other end (maximum pain score=10). The patients indicate the level of pain they perceive by pointing in accordance with their situation. The numerical data of the pain level of the individual is obtained by measuring the distance from the tip where there is no pain to the specified point with a ruler. The score is increased pain level increases. In the study conducted to ensure the standardization of the VAS, it is reported that the vertical use is better understood by the patients. The VAS has been used in many studies evaluating postoperative cesarean delivery pain. In this study, women's VAS scores were evaluated with a vertical form.

SECONDARY OUTCOMES:
Postpartum pain evaluation for abdomen | Since postpartum arrival to the clinic (postpartum hour 1) up to 48 hours
  Postpartum pain level evaluation for abdomen in this study is same the pain assessment postpartum cesarean section incision and is determined using VAS.
Puerperal bleeding amount measurement | Since postpartum arrival to the clinic (postpartum hour 1) up to 48 hours
  Puerperal bleeding amount is measured by subtracting the known dry weights (gr) of the pads from those with bleeding, using a sensitive electronic scale.
Postpartum hemoglobin level and hematocrit ratio | Up to postpartum 24th hours
  Postpartum hemoglobin level (g/dl) and hematocrit ratio (%) is obtained from the hospital records in the 6th and 24th hours.
Breastfeeding success evaluation | Since postpartum arrival to the clinic (postpartum hour 1) up to 48 hours
  Breastfeeding success is determined by using the Breastfeeding Assesment Scale [LATCH]. LATCH is similar to the APGAR scoring system and consists of 5 items:
  * L; how well the infant latches onto the breast,
  * A; audible/visible swallowing of the infant,
  * T; type of nipple,
  * C; mother's level of comfort regarding the breast and nipple, and
  * H; position for holding the baby. Each item of the scale is scored as 0, 1 or 2. The score range is 0 to 10. Higher total scores indicate higher success with breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Kara, MSc, Principal Investigator — Nigde Omer Halisdemir University; Evşen Nazik, PhD, Study Director — Cukurova University
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
This study will be published as a doctoral thesis. It is also planned to be published as a research article in a scientific journal.
Supporting Information: Study Protocol
Time Frame: 2 year
Access Criteria: The published protocol can be used to set an example for scientific research planning. The principal investigator can be contacted to provide data source for meta-analysis and systematic review studies.

REFERENCES:
- [Derived] Kara P, Nazik E. The effect of an abdominal binder on pain, bleeding and breastfeeding success after cesarean delivery: A randomized controlled trial. Women Health. 2025 Feb;65(2):124-139. doi: 10.1080/03630242.2024.2448514. Epub 2025 Jan 8. PMID 39780504